CLINICAL TRIAL: NCT01554228
Title: Change in Cognitive Function in Obese Patients After Bariatric Surgery - an Observational Study
Acronym: Obesity
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr. med. Agnes Floeel, Charite University, Berlin, Germany
Other Study IDs: Obes_Sur_Cog
Record Dates: First submitted 2012-03-13; First posted 2012-03-14 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric Surgery
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observational study to examine changes in cognition following bariatric surgery after one year.

SUMMARY:
Bariatric surgery provides a strong and long-term effect in reducing weight in obese subjects. Studies showed that obesity and its comorbidities are associated with a lower cognitive performance. The aim of the researchers study is to examine the cognitive performance of the patients before and after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* Age: 18-60

Exclusion Criteria:

* BMI < 40
* Age < 18 and > 60
* Presence of Cancer
* Presence of Chronic Inflammatory Diseases
* Presence of Addiction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients from the surgery department of the Charite Universtiy Berlin
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
performance in a neuropsychological test battery before and after surgery | 6 month

SECONDARY OUTCOMES:
performance in neuropsychological test battery 12 month after surgery compared to performance after 6 month and baseline performance | 12 month
performance in further cognitive tests | 6 - 12 month
surrogat parameters, blood parameters | 6-12 month

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof. MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Surgery Department, Charite University, Berlin, Germany